CLINICAL TRIAL: NCT04062968
Title: The Effect of Standardized Video Education on Prenatal Genetic Testing Choices, Decisional Conflict, and Decisional Regret
Brief Title: Video Education for Prenatal Testing Choices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Naval Medical Center, San Diego (U.S. Federal Agency)
Responsible Party: Principal Investigator, Monica Lutgendorf, Principal Investigator, United States Naval Medical Center, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NMCSD.2016.0070
Record Dates: First submitted 2019-08-07; First posted 2019-08-20 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Pregnancy

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to video education or usual care. Randomization will be completed using a random number table. Women randomized to the intervention group (video education) will view the prenatal screening video made by the Genetic Support Foundation and the Washington Department of Health, the 4.5 minute video "How to Decide About Prenatal Genetic Testing," available at: https://www.geneticsupportfoundation.org/genetics-and-you/pregnancy-and-genetics/prenatal-genetic-testing-videos .7 They will then complete the study related surveys at their initial obstetric visit.
  Women randomized to the control group will receive routine prenatal care with no additional study intervention other than completion of the study related surveys at baseline (initial prenatal testing).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video education (Experimental): Women randomized to the intervention group (video education) will view the prenatal screening video made by the Genetic Support Foundation and the Washington Department of Health, the 4.5 minute video "How to Decide About Prenatal Genetic Testing," available at: https://www.geneticsupportfoundation.org/genetics-and-you/pregnancy-and-genetics/prenatal-genetic-testing-videos .7 They will then complete the study related surveys at their initial obstetric visit.
  Interventions: Other: Video education
- Usual care (No Intervention): Women randomized to the control group will receive routine prenatal care with no additional study intervention other than completion of the study related surveys at baseline (initial prenatal testing).

INTERVENTIONS:
Other: Video education — Prenatal screening video made by the Genetic Support Foundation and the Washington Department of Health, the 4.5 minute video "How to Decide About Prenatal Genetic Testing," available at: https://www.geneticsupportfoundation.org/genetics-and-you/pregnancy-and-genetics/prenatal-genetic-testing-videos .
  Arms: Video education

SUMMARY:
The purpose of the investigator's study is to assess the effect of a standardized prenatal testing educational video on the use of prenatal genetic testing and decision-making.

DETAILED DESCRIPTION:
This is a prospective randomized trial of video education on prenatal testing vs. usual care, with the goal to assess women's prenatal testing choices, understanding of testing options and decisional conflict and regret. Participants will be recruited from a convenience sample of patients presenting for prenatal care at Naval Medical Center San Diego (NMCSD).

While receiving prenatal care at NMCSD, all women are offered the option of screening for aneuploidy (serum screen (with or without nuchal translucency ultrasound) or cell free DNA testing) or diagnostic testing (chorionic villous sampling or amniocentesis) or no testing in pregnancy.

After providing consent, participants will be randomized to video education or usual care. Randomization will be completed using a random number table. Women randomized to the intervention group (video education) will view the prenatal screening video made by the Genetic Support Foundation and the Washington Department of Health, the 4.5 minute video "How to Decide About Prenatal Genetic Testing," available at: https://www.geneticsupportfoundation.org/genetics-and-you/pregnancy-and-genetics/prenatal-genetic-testing-videos .7 They will then complete the study related surveys at their initial obstetric visit. The educational video was created with input from clinicians including licensed genetic counselors, obstetricians, maternal fetal medicine physicians, and patients. Extensive testing and reviewing was completed to ensure adequate comprehension by a wide range of audiences and minimize counseling bias. Women randomized to the control group will receive routine prenatal care with no additional study intervention other than completion of the study related surveys at baseline (initial prenatal testing). Current national guidelines recommend offering all women prenatal diagnosis and prenatal screening at the beginning of the pregnancy.1

The primary outcome for this study will be screening uptake rates, and will be based on review of the patient's electronic medical record. Secondary outcomes will include invasive diagnostic test rates, participant knowledge about testing (as assessed using the Maternal Serum Screening Knowledge Questionnaire,2 and decisional conflict (as assessed by the Decisional Conflict Scale) and decisional regret (as assessed by the Decision Regret Scale). These assessments will be conducted at time of prenatal testing (< 20 weeks). (Appendix A)

The study questionnaire will include a check box for participants to indicate if they would be willing to participate in a follow on qualitative study to assess participant's personal experience related to their method of education about prenatal testing. This component of the study will aim to determine personal and social reasoning behind their decisions, and to further explore their experience, beliefs and behaviors. Interested participants from each group (both intervention and control) will be contacted to arrange a telephone or in person interview. (Appendix C) Participants will be interviewed in person or over the phone.

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to 18 years of age
* Gestational age less than or equal to 20 weeks
* Singleton gestation
* Not completed aneuploidy screening in this pregnancy
* Available to watch the 15 minute video
* Ability to read, write, and understand English

Exclusion Criteria:

* Pregnant women not eligible for care at Military Treatment Facility
* Less than 18 years of age
* Gestational age greater than 20 weeks
* Multiple gestation
* Aneuploidy testing in current pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2017-01-12 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
screening uptake rates | 24-36 weeks gestation
  Genetic screening

SECONDARY OUTCOMES:
Invasive diagnostic test rates | 24-36 weeks gestation
  Diagnostic testing such as Chorinonic Villus Sampling and amniocentesis
Participant knowledge about prenatal testing | up to 20 weeks gestation
  Assessed by using the Maternal Serum Screening knowledge Questionnaire. Scores range from 0 to 15, reflecting the number of correct answers. A score of zero would indicate zero correct answers, where a score of 15 would indicate all answers were correct. Higher scores are considered better outcome indicating higher knowledge.
Decisional conflict | up to 20 weeks gestation
  Assessed by the Decisional Conflict Scale. Questions are scored on a Likert scale of 1 to 5, with 1 equating to Strongly Agree and 5 equating to Strongly Disagree. Thus, lower scores indicate lower decisional conflict. Subscale Decisional Uncertainty score range 3 to 15. Subscale Percieved Effective Decision range 4 to 20.
Decisonal regret | up to 20 weeks gestation
  Assessed by the Decisional Regret Scale. Questions are scored on a Likert scale of 1 to 5, with 1 equating to Strongly Agree and 5 equating to Strongly Disagree. Thus, lower scores indicate lower decisional regret. Decisional Regret scores range 0 to 100.

CONTACTS AND LOCATIONS:
Locations (1):
- Naval Medical Center San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No